CLINICAL TRIAL: NCT01064804
Title: An Open Randomised 4-Way Crossover Single Dose And A Parallel Group Multiple Dose Comparative Pharmacokinetic Study Of The PF-04191834 Phase 2 Tablet And The Phase 1 Dispersion Formulations.
Brief Title: To Test The Relative Bioavailability Of PF-04191834 When Dosed As An Immediate Release Tablet Compared With Solution Following Single And Multiple Dosing
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Other Study IDs: B0041005
Record Dates: First submitted 2009-09-01; First posted 2010-02-08 (Estimated); Last update posted 2010-02-08 (Estimated); Status verified 2010-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, plasma, urine, saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- relative bioavailability
  Interventions: Drug: PF-04191834

INTERVENTIONS:
Drug: PF-04191834 — PF-04191834. 100mg Immediate Release Tablets or oral suspension

SUMMARY:
To test the relative bioavailability of PF-04191834 when dosed as an Immediate Release tablet compared with solution following single and multiple dosing.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects between the ages of 18 and 55 years, inclusive (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG and clinical laboratory tests).
* Body Mass Index (BMI) of approximately 17.5 kg/m2 to 30.5 kg/m2 and a total body weight > 50 kg (110 lbs).
* An informed consent document signed and dated by the subject or a legally acceptable representative.
* Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
* Subjects who have urinary LTE4 levels greater than or equal to 30 pg/mg Creatinine at screening following spot urinary collection for Cohort 2.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Any condition possibly affecting drug absorption (eg, gastrectomy).
* A positive urine drug screen.

Ages: 21 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: young, healthy male volunteers
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2009-09; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
pharmacokinetic parameters of PF-04191834 | hours

SECONDARY OUTCOMES:
maximum concentration

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0041005&StudyName=To%20Test%20The%20Relative%20Bioavailability%20Of%20PF-04191834%20When%20Dosed%20As%20An%20Immediate%20Release%20Tablet%20Compared%20With%20Solution%20Following%20Single%20An